CLINICAL TRIAL: NCT03273374
Title: A Prospective, Phase II Study Investigating Efficacy of Intraoperative Radiation Therapy for Resectable Pancreatic Cancer
Brief Title: Intraoperative Radiation Therapy for Resectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Ik Jae Lee, Principal Investigator, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2017-0171
Record Dates: First submitted 2017-09-03; First posted 2017-09-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Resectable Pancreatic Adenocarcinoma

STUDY DESIGN:
Intervention Model Description: Intervention: intraoperative radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IORT group (Experimental): Intraoperative radiation therapy of 10 Gy delivered during surgery followed by adjuvant gemcitabine chemotherapy
  Interventions: Device: Intraoperative radiation therapy (IORT)

INTERVENTIONS:
Device: Intraoperative radiation therapy (IORT) — IORT with 50 kV x-ray will be delivered during surgery as a single dose of 10 Gy at 5 millimeter depths of the tumor bed, followed by gemcitabine chemotherapy (1000 mg/m2) every 4 weeks for a total of 6 cycles

SUMMARY:
This phase II study is designed to investigate the efficacy of IORT for patients with resectable pancreatic adenocarcinoma. The purpose of the study is to show the local recurrence rate after surgical resection and IORT is superior to that of surgical resection alone from the historical control. A total of 42 patients will be enrolled, and these patients will receive IORT of 10 Gy at 5 millimeter depth of the tumor bed, followed by 6 cycles of adjuvant gemcitabine chemotherapy.

DETAILED DESCRIPTION:
Treatment outcomes of pancreatic cancer are poor even after surgical resection, thus patients may receive adjuvant chemotherapy or chemoradiotherapy. Intraoperative radiotherapy (IORT) with low energy (50 kV) x-ray allows delivery of a high dose radiation to the tumor bed during surgery while effectively sparing adjacent critical organs. Another advantage of IORT is that delivery of IORT does not interfere with the scheduled administration of adjuvant chemotherapy or chemoradiotherapy. Here we investigate the efficacy of IORT for patients with resectable pancreatic adenocarcinoma by comparing the local recurrence rate after surical resection and IORT with that of surgical resection alone from the historical control. A total of 42 patients will be enrolled in this phase II trial, and these patients will receive IORT of 10 Gy at 5 millimeter depth of the tumor bed, followed by 6 cycles of adjuvant gemcitabine chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathologically confirmed pancreatic adenocarcinoma 2. Age ≥20 years 3. Performance status ECOG 0-2 4. Patients must have resectable disease. In order to be resectable the following criteria must be met:
* Absence of distant metastases
* Clear fat planes around the celiac axis, hepatic artery, and superior mesenteric artery
* Absence of direct involvement of inferior vena cava or aorta
* Stage I-III disease per AJCC 7th edition 5. Laboratory data obtained ≤14 days prior to registration on study, with adequate bone marrow and renal function defined as follows:
* Hemoglobin >10 g/dL, Absolute Neutrophil Count (ANC) >1,500/mm3, Platelets >100,000/mm3
* Serum Cr <1.4 mg/dL, BUN <20 mg/dL 6. Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* 1. Patients who have received external beam radiotherapy in the abdominal area 2. Defined treatment area which cannot be adequately covered by the radiation field as defined by the radiation oncology treatment team 3. Patients who have received neoadjuvant chemotherapy 4. Stage IV disease 5. Patients with distant metastases 6. Current pregnancy or currently nursing

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2020-08-21 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Local recurrence rate | 12 months
  Local recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: Ik Jae Lee, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho Y, Kim JW, Kim HS, Park JS, Lee IJ. Intraoperative Radiotherapy for Resectable Pancreatic Cancer Using a Low-Energy X-Ray Source: Postoperative Complications and Early Outcomes. Yonsei Med J. 2022 May;63(5):405-412. doi: 10.3349/ymj.2022.63.5.405. PMID 35512742
- [Derived] Lee YS, Kim HS, Cho Y, Lee IJ, Kim HJ, Lee DE, Kang HW, Park JS. Intraoperative radiation therapy induces immune response activity after pancreatic surgery. BMC Cancer. 2021 Oct 12;21(1):1097. doi: 10.1186/s12885-021-08807-3. PMID 34641806
- [Derived] Kim JW, Cho Y, Kim HS, Choi WH, Park JS, Lee IJ. A phase II study of intraoperative radiotherapy using a low-energy x-ray source for resectable pancreatic cancer: a study protocol. BMC Surg. 2019 Mar 7;19(1):31. doi: 10.1186/s12893-019-0492-x. PMID 30845939